CLINICAL TRIAL: NCT04794218
Title: A Phase 1 Randomized, Double-blinded, Placebo-controlled, Dose-escalation Clinical Trial to Evaluate the Safety and Immunogenicity of rVSV∆G-LASV-GPC Vaccine in Adults in Good General Heath
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of rVSV∆G-LASV-GPC Vaccine in Adults in Good General Heath
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: George Washington University (Other); Brigham and Women's Hospital (Other); Redemption Hospital (Unknown); East-West Medical Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IAVI C102
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Lassa Fever; Lassa Virus Infection
MeSH Terms: conditions — Lassa Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Study Group 1 (Experimental): rVSV∆G-LASV-GPC Vaccine Dosage (pfu) intramuscularly Day 1 2 X 10^4 or Placebo
  Interventions: Drug: rVSV∆G-LASV-GPC; Other: Placebo/Diluent
- Study Group 2 (Experimental): rVSV∆G-LASV-GPC Vaccine Dosage (pfu) intramuscularly Day 1 2 X 10^5 or Placebo
  Interventions: Drug: rVSV∆G-LASV-GPC; Other: Placebo/Diluent
- Study Group 3 (Experimental): rVSV∆G-LASV-GPC Vaccine Dosage (pfu) intramuscularly Day 1 2 X 10^6 or Placebo
  Interventions: Drug: rVSV∆G-LASV-GPC; Other: Placebo/Diluent
- Study Group 4A (Experimental): rVSV∆G-LASV-GPC Vaccine Dosage (pfu) intramuscularly Day 1 2 X 10^7 or Placebo
  Interventions: Drug: rVSV∆G-LASV-GPC; Other: Placebo/Diluent
- Study Group 5 (Experimental): rVSV∆G-LASV-GPC Vaccine Dosage (pfu) intramuscularly Day 1 2 X 10^5 or Placebo
  Interventions: Drug: rVSV∆G-LASV-GPC; Other: Placebo/Diluent
- Study Group 6 (Experimental): rVSV∆G-LASV-GPC Vaccine Dosage (pfu) intramuscularly Day 1 2 X 10^6 or Placebo
  Interventions: Drug: rVSV∆G-LASV-GPC; Other: Placebo/Diluent
- Study Group 7 (Experimental): rVSV∆G-LASV-GPC Vaccine Dosage (pfu) intramuscularly Day 1 2 X 10^7 or Placebo
  Interventions: Drug: rVSV∆G-LASV-GPC; Other: Placebo/Diluent
- Study Group 4B (Experimental): rVSV∆G-LASV-GPC Vaccine Dosage (pfu) intramuscularly Day 1 and Day 42 2 X 10^7 or Placebo
  Interventions: Drug: rVSV∆G-LASV-GPC; Other: Placebo/Diluent

INTERVENTIONS:
Drug: rVSV∆G-LASV-GPC — 2 × 10^4 pfu delivered intramuscularly
  Arms: Study Group 1
Drug: rVSV∆G-LASV-GPC — 2 × 10^5 pfu delivered intramuscularly
  Arms: Study Group 2; Study Group 5
Drug: rVSV∆G-LASV-GPC — 2 × 10^6 pfu delivered intramuscularly
  Arms: Study Group 3; Study Group 6
Drug: rVSV∆G-LASV-GPC — 2 × 10^7 pfu delivered intramuscularly
  Arms: Study Group 4A; Study Group 4B; Study Group 7
Other: Placebo/Diluent — N/A delivered intramuscularly

SUMMARY:
A Phase 1 Randomized, Double-blinded, Placebo-controlled, Dose-escalation Clinical Trial to Evaluate the Safety and Immunogenicity of rVSV∆G-LASV-GPC Vaccine in Adults in Good General Health

DETAILED DESCRIPTION:
This is a Phase 1 Randomized, Double-blinded, Placebo-controlled, Dose-escalation Clinical Trial to Evaluate the Safety and Immunogenicity of rVSV∆G-LASV-GPC Vaccine in Adults in Good General Health.

Approximately 110 participants (88 active product and 22 placebo recipients) will be included in the study Participants will be screened up to 42 days before IP administration and will be followed for 12 months after IP administration.

ELIGIBILITY:
Inclusion Criteria

1. Adults in good general health as assessed by medical history, physical examination, and laboratory tests
2. At least 18 years of age on the day of screening and has not reached his/her 51st birthday on the day of vaccination
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study
4. Willing to undergo HIV testing, risk reduction counselling, and receive HIV test results
5. Use effective method of contraception
6. Understand the study and provide written informed consent

Exclusion Criteria

1. Confirmed HIV-1 or HIV-2 infection
2. Any clinically relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease
3. Any clinically significant chronic medical condition that, in the opinion of the Investigator, makes the participant unsuitable for participation in the study
4. Pregnant or lactating
5. Bleeding disorder that was diagnosed by a physician
6. Prior receipt of another investigational Lassa vaccine candidate
7. Receipt of blood transfusion or blood-derived products within the previous 3 months
8. Prior exposure to LASV as documented by history
9. History of severe local or systemic reactogenicity to any vaccine
10. Body mass index (BMI) ≥35
11. Mild or greater hearing impairment defined as ≥26dB loss in either ear

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Safety: To evaluate the safety and tolerability of rVSV∆G-LASV-GPC vaccine | 20 months
  * Proportion of participants with Grade 3 or higher reactogenicity (ie, solicited AEs) during a 14-day follow-up period after IP administration
  * Proportion of participants with Grade 2 or higher IP-related unsolicited AEs, including safety laboratory parameters, within 28 days of IP administration
  * Proportion of participants with Grade 2 or higher unsolicited AEs, including safety laboratory parameters, within 28 days of IP administration
  * Proportion of participants with IP-related SAEs throughout the study period Proportion of participants with AEs of Special Interest (AESI) post-vaccination throughout the study period

SECONDARY OUTCOMES:
Immunogenicity: To determine LASV-GPC-specific antibody responses induced by rVSV∆G-LASV-GPC vaccine | 20 months
  * Magnitude and duration of viral RNA in plasma by PCR
  * Magnitude and duration of rVSV∆G-LASV-GPC vaccine viremia by culture
  * Magnitude and duration of viral RNA in urine and saliva by PCR
  * Magnitude and duration of rVSV∆G-LASV-GPC vaccine shedding in urine and saliva by culture

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - George Washington University, Washington D.C., District of Columbia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Brigham and Women's Hospital, Brookline, Massachusetts
- Redemption Hospital, New Kru Town, Greater Monrovia, Liberia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malkin E, Zaric M, Kieh M, Baden LR, Fitz-Patrick D, Marini A, Yun H, Hayes P, Bromell R, Ayorinde M, Fernandez N, Varma R, Sigei F, Ward M, Pindolia H, Sewell S, Amini F, Blie J, Wilson B, Faley P, McCullough J, Tokpah F, Wisseh C, Towalid E, Hadawale S, Sayeed E, Hunt D, Keshavarzi N, Barin B, Maljkovic Berry I, Parks CL, Truter SG, Walker K, Vekemans J, Lehrman J, Engelbrecht M, Malherbe M, Laufer D, Philiponis V, Higgs E, Mutua G, Fast PE, Gupta SB; rVSVDeltaG-LASV-GPC Study Group. Safety and Immunogenicity of an rVSV Lassa Fever Vaccine Candidate. N Engl J Med. 2025 Nov 6;393(18):1807-1818. doi: 10.1056/NEJMoa2501073. PMID 41191941
- See also: Related Info — https://www.iavi.org/